CLINICAL TRIAL: NCT06212388
Title: Efficacy and Safety of Allogeneic γδ T Cells (γδ T Cells) Combined With Interferon-alpha1b (IFN-α1b) or PD-1 Monoclonal Antibody in Neoadjuvant Treatment of Stage III-IV Resectable Melanoma
Brief Title: Allogeneic Gammadelta T Cells Combined With Interferon-α1b or PD-1 Monoclonal Antibody in Stage III-IV Amenable to Surgical Resection Melanoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Beijing GD Initiative Cell Therapy Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDT-001-08
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: IFN-α1B+ γδ T cells (Experimental): Stage 1: Neoadjuvant stage (Week 1-9, 3 cycles)
  Stage 2: Surgical period (2 weeks, ±7 days after the last dose of neoadjuvant therapy) After multidisciplinary MDT team evaluation, the primary lesion and metastasis were resected in the corresponding departments.
  Stage 3: Postoperative adjuvant period (3 weeks ±7 days -45 weeks, 15 cycles) γδ T cells administered intravenously every three weeks. Recombinant human interferon α1b administered 300μg every other day.
  Interventions: Biological: Ex-vivo expanded allogeneic γδ T cells; Drug: Recombinant human interferon α1b
- group B: Palizizumab+ γδ T cells (Active Comparator): Stage 1: Neoadjuvant stage (Week 1-9, 3 cycles)
  Stage 2: Surgical period (2 weeks, ±7 days after the last dose of neoadjuvant therapy) After multidisciplinary MDT team evaluation, the primary lesion and metastasis were resected in the corresponding departments.
  Stage 3: Postoperative adjuvant period (3 weeks ±7 days -45 weeks, 15 cycles) γδ T cells administered intravenously every three weeks.Pembrolizumab administered 200mg intravenously every three weeks.
  Interventions: Biological: Ex-vivo expanded allogeneic γδ T cells; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Ex-vivo expanded allogeneic γδ T cells — Cells will be extracted from a healthy donor by apheresis, followed by ex-vivo expansion and activation. The ex-vivo expanded γδT cells from donors will be adoptively transfused.
Drug: Recombinant human interferon α1b — Recombinant human interferon α1b is a protein with potent antiviral, antiproliferative and immunomodulatory properties.
  Arms: group A: IFN-α1B+ γδ T cells
Drug: Pembrolizumab — Pembrolizumab is a recombinant, humanized programmed death receptor (PD-1) monoclonal antibody that binds to PD- and prevents binding of PD-1 with programed death ligands 1 (PD-L1) and PD-L2. It can function to activate cytotoxic T lymphocytes and inhibit tumor growth.
  Arms: group B: Palizizumab+ γδ T cells

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of allogeneic γδ T cells combined with recombinant human interferon-α1b (IFN-α1b) or PD-1 monoclonal antibody in neoadjuvant treatment of patients with Stage III-IV resectable melanoma.

DETAILED DESCRIPTION:
This is a double-arm, single-center, randomized, open label Phase I clinical trial to evaluate the efficacy and safety of the combination of ex-vivo expanded allogeneic γδ T cells plus recombinant human interferon α1b or PD-1 monoclonal antibody in patients with Stage III-IV resectable melanoma(AJCC 8th). We randomly assigned patients with stage III-IV melanoma that was amenable to surgical resection to three doses of neoadjuvant γδT cells plus IFN-α1b or γδT cells plus pembrolizumab , surgery, and 15 doses of adjuvant γδT cells plus IFN-α1b or γδT cells plus pembrolizumab. The primary endpoints are pathological response rate after 3 cycles of treatment, including: complete pathological response rate (pCR), major pathological response rate (MPR), partial pathological response rate (pPR); preoperative imaging response rate (RECIST v1.1) was evaluated, including complete response (CR), partial response (PR), stable disease (SD), and disease progression (PD); and proportion of patients who do not need surgery due to remission. The second endpoints are event-free survival (EFS), relapse free survival (RFS), and overall survival (OS, 3 years after surgery). The safety profile of the combined γδT cells/IFN-α1b regimen and γδT cells/ pembrolizumab regimen will be monitored, we will evaluate the numbers and severity of toxicity per the Criteria for Adverse Events version 5 (CTCAEv) including but not limited to all adverse events (AE), incidence of surgery-related adverse events, and proportion of inoperable patients (due to disease progression or treatment-related adverse events).

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75. 2. ECOG performance status of 0 or 1 3. Life expectancy ≥ 3 months; 4. Histologically or cytologically confirmed diagnosis of resectable stage III-IV melanoma by the American Joint Committee on Cancer (AJCC) (the 8th Edition). (Note: uveal melanoma cases are excluded) 5. Adequate organ and marrow function (within 4 weeks prior to study treatment initiation): 6. A negative urine or plasma β-HCG test result is required at screening for female patients of childbearing potential.

  7. Contraception is required for patients and their partners throughout the trial and within 1 year after the last dose of study treatment.

  8. Capable of understanding and complying with the study protocol requirements ( including follow-up visit and examinations).

  9. Be willing to signed a written informed consent document before enrollment.

Exclusion Criteria:

* 1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ex-vivo expanded allogeneic γδ T cells, recombinant human interferon-α1b and PD-1 monoclonal antibody.

  2. Patients accepted other anti-tumor clinical trials within 4 weeks prior to study entry.

  3. Patients accepted anti-tumor radiotherapy within 4 weeks prior to study entry.

  4. Disease improved by in response to anti-tumor therapies within 4 weeks including perioperative chemotherapy, molecularly targeted therapy, PD-1/PD-L1/CTLA-4 immune therapy, anti-angiogenesis therapy, interferon, herbal supplements, and other cell therapies including NK, CIK, DC, CTL and stem cell therapy etc.

  5. Plan to take other systemic or local anti-tumor therapy during the current study 6. Systemic treatment with either corticosteroid (> 10 mg /kg prednisone equivalents) or other immunosuppressive medications prior to 2 weeks prior to study dose initiation 7. Known hematologic malignancy, primary brain tumor, sarcoma or any other primary solid tumor unless the disease-free period is over 5 years.

  8. Imaging confirmed of central nervous system (CNS) metastases with or without meningeal carcinomatosis 9. Known severe hypersensitivity reaction of another adoptive immune cell therapy.

  10. Known active autoimmune disease requiring systemic treatment (such as corticosteroids or immunosuppressive medications) or related replacement therapies (such as thyroid hormone for hypothyroidism, insulin for diabetes or physiological glucocorticoid replacement therapy for adrenal or pituitary insufficiency) in the past 2 years.

  11. Surgery history within past 4 weeks, except for melanoma removal or partial removal.

  12. Major organs dysfunction. 13. Acute infections and any condition has potential risk of gastrointestinal bleeding or perforation, such as active gastrointestinal ulcer, known intra luminal metastases,inflammatory bowel disease; known abdominal fistula, gastrointestinal perforation or intraperitoneal abscess 4 weeks prior to entry of the study entry.

  14. Other diseases that may affect compliance or interfere with results interpretation including active opportunistic infections or progressing or severe infections , uncontrolled diabetes or pulmonary diseases including interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm.

  15. Known HIV or AIDS-related illness, or active HBV, HCV and tuberculosis. 16. A history of getting a live vaccine within 4 weeks prior to the first dose; a history of hematopoietic stimulating factor therapy such as colony-stimulating factor (CSF) and erythropoietin (EPO) within 2 weeks prior to the first dose; a history of major surgeon except for diagnosis within 4 weeks prior to the first dose.

  17. Diagnosis of a psychiatric or substance abuse disorder. 18. Individuals who are pregnant or breast-feeding or plan to conceive during the study period 19. Any other illness, laboratory abnormality, or situations that in the opinion of the principal investigator would compromise the patients' ability to tolerate treatment or would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-24 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Pathological Complete Response (pCR) | at 12 weeks
  Investigators will measure the rate of pCR after surgery.
Rate of Major Pathological Response (mPR) | at 12 weeks
  Investigators will measure the rate of mPR after surgery.
Rate of Partial Pathological Response (pPR) | at 12 weeks
  Investigators will measure the rate of pPR after surgery.
Overall Response Rate(ORR) | up to 12 weeks
  ORR will be measured after neoadjuvant therapy (for participants who have measurable disease per RECIST 1.1 at start of neoadjuvant therapy).

SECONDARY OUTCOMES:
Event Free survival(EFS) | From randomization up to 3 years after surgery
  EFS is defined as time from randomization to melanoma progression (irresectable stage III or stage IV disease), melanoma recurrence, treatment-related death, or melanoma-related death, whichever occurs first. Occurrence of a new primary melanoma during treatment/follow-up is also regarded as an event. Presurgical resectable progression to stage III disease is not defined as an event, even as death to another reason than melanoma or the study treatment.
Relapse Free Survival (RFS) | After surgery up to 3 years
  RFS is defined as time from surgery until disease relapse.
3 Year Overall Survival (OS) | After surgery up to 3 years
  The 3 years after surgery OS rate of patients with γδ T cells plus IFN-α1B or γδ T cells plus pembrolizumab，From date of enrollment until the date of death from any cause.
Incidence of Adverse Events (AEs) | After surgery up to 13 months
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

IPD SHARING:
Plan to Share IPD: No